CLINICAL TRIAL: NCT06145672
Title: Definitive Treatment of Alopecic Scars by Follicular Unit Extraction Hair Transplantation, Randomized Prospective Controlled Study
Brief Title: Treatment of Alopecic Scars by Follicular Unit Extraction Hair Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maged Medhat Armaneous, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Follicular Unit Extraction
Record Dates: First submitted 2023-10-26; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Alopecia Scar
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: To hide alopecic scars with some hairs harvested as FUs at the back of the scalp under local anaesthesia without leaving any residual deformity or adding more scars to the donor area and implant it in the non-hairy scars.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mature Alopecic Scars (Active Comparator): Follicular Unit Extraction and implantation for Alopecic Scars in beard Follicular Unit Extraction and implantation for Alopecic Scars in scalp Follicular Unit Extraction and implantation for Alopecic Scars in eyebrow Follicular Unit Extraction and implantation for Alopecic Scars in Moustache
  Interventions: Procedure: follicular unit extraction and implantaion
- Immature Alopecic Scars (Experimental): Follicular Unit Extraction and implantation for Alopecic Scars in beard Follicular Unit Extraction and implantation for Alopecic Scars in scalp Follicular Unit Extraction and implantation for Alopecic Scars in eyebrow Follicular Unit Extraction and implantation for Alopecic Scars in Moustache
  Interventions: Procedure: follicular unit extraction and implantaion

INTERVENTIONS:
Procedure: follicular unit extraction and implantaion — extract hair follicles as grafts from donor area and implant them in recipient area

SUMMARY:
This study aim: is to completely hide the alopecic scars in a way that it will not be visible.

DETAILED DESCRIPTION:
Practicing scar revision, there is an increasing demand for almost complete reconstruction and camouflaging scars in hairy areas rather than scars in non-hairy skin. Scar revision rendered insufficient reconstructive tool in such cases. Whatever a Plastic surgeon pay efforts in alopecic scars rejuvenation and reconstruction, it is still apparent and noticeable. One of the best surgical techniques to camouflage an alopecic scar is hair transplantation. FUE is the state-of-the-art technique for hair transplantation.

In the field of hair restoration, there has been a significant increase in demand with patients for facial hair transplantation procedures. Modern techniques in hair transplantation is based on follicular unit extraction and implantation, in which follicular units are the exclusive structures used as hair grafts allow for facial hair transplantation and for the attainment of natural-appearing results. Facial hair transplantation is a subspecialty within hair restoration with many gratifying benefits for the patients as well as for the hair restoration surgeon. Adapting these advanced techniques into a hair restoration practice allows a surgeon to offer their patients these procedures and provides an expanded artistic element to a hair restoration surgeon's practice. The art and science of hair transplantation have come a long way since its introduction in 1959. Both the technique and instruments have been greatly improved, thus offering the patient an excellent cosmetic result that will last a lifetime.

ELIGIBILITY:
Inclusion Criteria:

* small scalp alopecic scars.
* post traumatic alopecic beard scars
* post traumatic alopecic moustache scars.
* post traumatic alopecic scalp scars.
* post traumatic alopecic eyebrow scars.
* post burn small alopecic scars.
* mature scars.
* controlled infective scars.

Exclusion Criteria:

* large alopecic scars
* post burn alaopecic scar
* uncontrolled active scar
* male pattern baldness
* female pattern baldness

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
evaluating post operative pain using questionnaire | 6 Month - 1 year
  assessment of post operative pain and complications using questionnaire
evaluating post operative complications | 6 Month - 1 year
  assessment of post operative pain and complications using questionnaire
donor and recipient site assessment | 6 Month - 1 year
  care for recipient as well as donor site using questionnaire

SECONDARY OUTCOMES:
Follicular unit growth monitoring | monthly up to 1 year
  close monitoring for growth of FU growth
platlet rich plasma injection for FU growth | every 2 weeks up to 6 months
number of hairs in each hair follicle | every 2 weeks up to 3months

CONTACTS AND LOCATIONS:
Overall Officials: wael saadeldeen saadeldin, MD, Study Chair — Department of Plastic Surgery,

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jimenez F, Alam M, Vogel JE, Avram M. Hair transplantation: Basic overview. J Am Acad Dermatol. 2021 Oct;85(4):803-814. doi: 10.1016/j.jaad.2021.03.124. Epub 2021 Apr 24. PMID 33905785
- [Result] Bared A. Beard Hair Transplantation. Facial Plast Surg Clin North Am. 2020 May;28(2):237-241. doi: 10.1016/j.fsc.2020.01.010. PMID 32312510
- [Result] Pinski JB. Hair transplantation and bald-scalp reduction. Dermatol Clin. 1991 Jan;9(1):151-68. PMID 2022091
- [Result] Barreto OC. [Hair transplantation. Past, present, and future]. Acta Med Port. 1998 Mar;11(3):283-5. Portuguese. PMID 9741133
- [Result] Bernstein RM, Rassman WR. The logic of follicular unit transplantation. Dermatol Clin. 1999 Apr;17(2):277-95, viii; discussion 296. doi: 10.1016/s0733-8635(05)70087-5. PMID 10327298
- [Result] Bernstein RM, Rassman WR. Follicular transplantation. Patient evaluation and surgical planning. Dermatol Surg. 1997 Sep;23(9):771-84; discussion 801-5. PMID 9311372
- [Result] Chen L, Wang B, Liu X, Yang J, Jiang W. Comparison of 2 Incisional Methods in Hair Transplantation. J Craniofac Surg. 2023 Jul-Aug 01;34(5):e499-e501. doi: 10.1097/SCS.0000000000009372. Epub 2023 Jun 12. PMID 37307246